THYROID CANCER IN SURGICALLY TREATED

MULTINODULAR GOITER: INCIDENCE AND

HISTOPATHOLOGICAL OUTCOMES

NCT NUMBER not available.

Date of document: 15/12/2023

# **ABSTRACT**

### INTRODUCTION

Thyroid cancer, the most common endocrine malignancy, has been extensively studied due to its rising global incidence and diverse clinical presentations. Among thyroid disorders, multinodular goiter (MNG) is frequently encountered in clinical practice, with a prevalence ranging from 0.4% to 7.2% in iodine-sufficient regions and affecting approximately 25–33% of the population in iodine-deficient areas.

The association between MNG and thyroid cancer is well-documented, although reported incidence rates vary significantly among studies and populations, ranging from 5% to 35% in the literature This study aims to investigate, based on existing knowledge, the incidence of occult thyroid carcinoma in a cohort of patients with MNG, providing new insights into the prevalence and characteristics of thyroid malignancies in MNG. It seeks to contribute to optimizing diagnostic evaluations for patients with multinodular goiter.

### MATHERIALS AND METHODS

This retrospective study included patients with a preoperative diagnosis of multinodular goiter who underwent total or partial thyroidectomy from January 2018 to May 2024 at the Department of Medical and Surgical Sciences at the University Hospital "Ospedali Riuniti" in Foggia. The study's objective was to investigate the incidence of thyroid carcinoma in patients undergoing thyroidectomy for MNG, also analyzing associated demographic and clinical variables.

### **RESULTS**

Out of the 223 patients, 32 cases of thyroid carcinoma were diagnosed, corresponding to an incidence rate of 14.4%. Among these, 24 were female (75%) and 8 were male (25%), with a female-to-male

ratio of 3:1. Thyroid carcinoma was identified in 13.3% of all females and 19% of all males. Although a difference in incidence between the sexes was observed, it was not statistically significant (chi=0.929; p=0.335).

Papillary thyroid carcinoma (PTC) was the most common type, identified in 25 cases (78.1%).

The mean age of patients with thyroid carcinoma was 49.4 years (SD 16.7), with an age range of 22 to 72 years. A significant difference was observed between this group and the mean age of patients without carcinoma (mean: 56.2 years, SD 13.1). Statistical analysis indicated a significant difference between the two groups in terms of age (t=-2.686; p=0.008). Additionally, evaluating the correlation between age and malignancy revealed that for each additional year of age, the probability of carcinoma decreased by 3.7% (OR=0.963; p=0.009).

### CONCLUSION

The results of this study highlight a significant incidence of thyroid carcinoma in patients with multinodular goiter. The predominant histotype was papillary carcinoma, with no observed sex-based differences in incidence. The identified risk factors, such as age and thyroid weight, while potentially useful for stratifying risk in patients with multinodular goiter, are insufficient—due to study limitations and the significant variability among populations from different regions—to justify modifications to existing thyroid nodule screening criteria.

Keywords: multinodular goiter; incidental thyroid cancer; total thyroidectomy; endocrine surgery Introduction

Thyroid cancer, the most common endocrine malignancy, has been extensively studied due to its rising global incidence and diverse clinical presentations. Among thyroid disorders, multinodular goiter (MNG) is frequently encountered in clinical practice, with a prevalence ranging from 0.4% to 7.2% in iodine-sufficient regions and affecting approximately 25–33% of the population in iodine-deficient areas. [1] It is characterized by an enlarged thyroid gland containing multiple nodules. The pathogenesis of MNG involves various genetic, environmental, and dietary factors leading to the development of multiple thyroid nodules.

The association between MNG and thyroid cancer is well-documented, although reported incidence rates vary significantly among studies and populations, ranging from 5% to 35% in the literature [2]. Bove et al. reported an overall incidence of 8.9% in 2023, including 6.1% microcarcinoma cases and 2.8% thyroid carcinoma cases [3]. In 2021, a study involving 3,233 patients found thyroid carcinoma in 1,026 of them, corresponding to an incidence of 31.7% [4-5]. Another study conducted in Southern Italy, focusing on a genetically homogeneous population in Calabria with mild to moderate iodine deficiency, reported an overall prevalence rate of incidental thyroid carcinoma of 12.5% [6].

These differences may partially stem from genetic variability among populations and sociocultural factors, particularly diet. However, the relationship between iodine intake and thyroid cancer remains controversial. After iodine intake increased due to salt iodization and iodine supplementation, the incidence of thyroid cancer, particularly papillary thyroid carcinoma (PTC), rose despite a decrease in follicular thyroid carcinoma (FTC) incidence. Conversely, some meta-analyses on the association between iodine intake and thyroid cancer have found that higher iodine intake correlates with a lower risk of thyroid cancer [7]. Other studies indicate an association between excessive body fat, obesity, and overweight status with thyroid neoplasia [8; 9]. These findings highlight the intricate relationship between diet and thyroid pathology, emphasizing the need for optimal dietary strategies.

Although most nodules in MNG are benign, the presence of multiple nodules complicates the identification of potentially malignant ones. It has long been believed that the risk of cancer in MNG is much lower than in solitary nodules. However, recent literature indicates that if a nodule in MNG

grows consistently, becomes markedly dominant, or changes in consistency, its risk of malignancy matches that of a solitary nodule. Fineneedle aspiration (FNA) can differentiate thyroid nodules with a high risk of malignancy, warranting surgical removal, from benign goitrous nodules manageable with pharmacological therapy. FNA is associated with falsenegative rates of approximately 3% for solitary nodules [9]. However, the diagnostic process is complicated by the number of nodules and the need to select those for biopsy, which may reduce the sensitivity of the procedure [10-11]. The application of TIRADS ultrasound criteria can aid in identifying suspicious nodules, guiding further diagnostic assessments.

Advancements in molecular testing have also contributed to evaluating thyroid nodules. Nikiforov et al. (2011) discussed the use of molecular markers such as BRAF, RAS mutations, and RET/PTC rearrangements in predicting thyroid cancer. Their study demonstrated that integrating molecular testing with traditional diagnostic methods improves malignancy detection accuracy in MNG [12]. Similarly, Agrawal et al. (2012) highlighted the potential of molecular diagnostics to refine risk stratification and management of thyroid nodules [13].

The association between gender and thyroid cancer has yielded conflicting results. A recent study found that men had a higher risk of incidental papillary thyroid carcinoma [4], whereas others reported a higher prevalence of incidental thyroid carcinoma in the female population [3; 6].

The collective findings from these studies underscore the complex and only partially understood interaction between MNG and thyroid cancer. Although the incidence of malignancy within MNG is relatively low, a rigorous diagnostic approach is essential for the timely and accurate identification of tumors. Integrating ultrasound imaging, FNA, and molecular tests has enhanced diagnostic precision, enabling more informed clinical decisions. Moreover, identifying correlations with demographic and clinical factors could help refine risk stratification and patient management in MNG.

This study aims to investigate, based on existing knowledge, the incidence of occult thyroid carcinoma in a cohort of patients with MNG, providing new insights into the prevalence and characteristics of thyroid malignancies in MNG. It seeks to contribute to optimizing diagnostic evaluations for patients with multinodular goiter.

#### Materials and Methods

#### **Patients**

This retrospective study included patients with a preoperative diagnosis of multinodular goiter who underwent total or partial thyroidectomy from January 2018 to May 2024 at the Department of Medical and Surgical Sciences at the University Hospital "Ospedali Riuniti" in Foggia. The study's objective was to investigate the incidence of thyroid carcinoma in patients undergoing thyroidectomy for MNG, also analyzing associated demographic and clinical variables.

Diagnoses of multinodular goiter were confirmed through clinical and ultrasound examinations. Tissue samples obtained during surgery were analyzed by expert pathologists to identify thyroid carcinoma.

Inclusion criteria were: (1) patients diagnosed with multinodular goiter via thyroid ultrasound, with or without FNA cytology, (2) patients who underwent surgery, and (3) availability of complete clinical data. Exclusion criteria were: patients with a history of thyroid carcinoma or other thyroid neoplasms, those who did not complete postoperative follow up, and patients with preoperative FNA results indicating malignancy (TIR 4–5), suspicion of malignancy (TIR 3), or indeterminate significance (TIR 1) per the 2014 criteria of the Italian Society of Pathological Anatomy and Cytology (SIAPEC).

Demographic, clinical, and pathological data were collected from paper and/or electronic medical records. These included age, sex, results of any FNA cytology, type of surgery, weight of the resected thyroid, and definitive histopathological findings.

#### Statistical Analysis

Continuous variables were represented as mean values along with standard deviation (SD), while categorical variables were presented as counts and percentages. Percentages were compared using Pearson's chi-square test, a statistical method employed to assess whether the observed frequency distribution differs significantly from the expected distribution in a given sample. In essence, it evaluates whether two categorical variables are independent.

To investigate potential correlations between continuous variables and the presence of malignancy, an independent samples Student's t-test was conducted. This test determines whether there are statistically significant differences between the means of two groups.

Logistic regression analysis was performed to examine the potential relationship between age and incidental thyroid carcinoma (ITC). Logistic regression is a statistical test used to analyze the relationship between a binary dependent variable (e.g., yes/no, 0/1) and one or more independent variables. This method estimates the impact of independent variables on the dependent variable. The resulting odds ratios (OR) were reported with 95% confidence intervals (CI). A significance level of 0.05 was selected to determine statistical significance. Statistical analysis was conducted using SPSS software.

### Results

| Charateristics | Mean (SD) or Number (%) |
|-----------------------|-------------------------|
| Male, nº | 42 (18,8%) |
| Female, nº | 181 (81,2%) |
| Age, years | 55,3 (±13,5) |
| Benign FNA (TIR2), nº | 151 (67,7%) |
| FNA not done, n° | 72 (32,3%) |

Total thyroidectomy, n° 202 (90,6%)

Lobectomy, n° 21 (9,4%)

Thyroid wheight, grams 68,4 (±57,9)

Table 1: carateristics of the study partecipants

The study included a cohort of 223 patients diagnosed with multinodular goiter (MNG) at our center between January 2018 and May 2024. The cohort consisted of 181 females (81.2%) and 42 males (18.8%), with a mean age of 55.3 years (SD 15.5). All cases were benign multinodular goiter, with 151 patients (67.7%) undergoing fine-needle aspiration (FNA) yielding benign results, and 72 patients (32.3%) not undergoing FNA. All patients underwent surgical treatment for symptomatic goiter (compressive symptoms, hypo-/hyperthyroidism), with 202 (90.6%) undergoing total thyroidectomy and 21 (9.4%) undergoing lobectomy (Table 1). Patients diagnosed with incidental carcinoma post-total thyroidectomy were referred directly for endocrinological and oncological follow-up, while those who underwent lobectomy received the same guidance following completion of thyroidectomy.

| Charateristics | Mean (SD) or Number (%) |
|-------------------------|-------------------------|
| Carcinoma, nº | 32 (14,4%) |
| M | 8 (25%) |
| F | 24 (75%) |
| Benigne neoplasms, nº | 22 (10,9%) |
| Age, years | 49,4 (±16,7) |
| Benign FNA (TIR2), n° | 18 (56,3%) |
| FNA not done, n° | 18 (56,3%) |
| Total thyroidectomy, nº | 29 (90,6%) |
| Lobectomy, n° | 3 (9,4%) |
| Thyroide weight, grams | 50,9 (±48,1) |

Table 2: charateristics of patient with carcinoma

Out of the 223 patients, 32 cases of thyroid carcinoma were diagnosed, corresponding to an incidence rate of 14.4% (Table 2). Among these, 24 were female (75%) and 8 were male (25%), with a female-to-male ratio of 3:1. Thyroid carcinoma was identified in 13.3% of all females and 19% of all males. Although a difference in incidence between the sexes was observed, it was not statistically significant (chi=0.929; p=0.335).

The diagnosis of carcinoma was confirmed through postoperative histopathological examination, which classified the subtypes of thyroid carcinoma present in the sample. Papillary thyroid carcinoma (PTC) was the most common type, identified in 25 cases (78.1%), including 16 cases (50%) of microcarcinoma (pT1a; <1 cm) and 9 cases of classic PTC. Follicular thyroid carcinoma was diagnosed

in 5 cases (15.6%), while 1 case of anaplastic carcinoma and 1 case of Hurthle cell carcinoma were identified.





Figure 1: subtypes of thyroid carcinoma

Regarding benign neoplasms, 20 follicular adenomas, 1 Hurthle cell adenoma, and 1 NIFTP (non-invasive follicular thyroid neoplasm with papillary-like nuclear features) were identified.

The mean age of patients with thyroid carcinoma was 49.4 years (SD 16.7), with an age range of 22 to 72 years. A significant difference was observed between this group and the mean age of patients without carcinoma (mean: 56.2 years, SD 13.1; Figure 2). Statistical analysis indicated a significant difference between the two groups in terms of age (t=-2.686; p=0.008). Additionally, evaluating the correlation between age and malignancy revealed that for each additional year of age, the probability of carcinoma decreased by 3.7% (OR=0.963; p=0.009).



Figure 2: age in the groups whit an without carcinoma

No significant differences were found between the mean ages of male and female patients with carcinoma.

Following surgical removal, the weight of the thyroid glands was assessed as an indicative parameter of size, volume, and the density of the thyroid parenchyma, serving as a characteristic that integrates multiple structural factors of the organ affected by MNG.



Figure 3: weight in the groups with and without carcinoma

The mean thyroid weight in patients with ITC was 50.9 grams (SD 48.1), compared to 71.3 grams (SD 59.0) in patients without ITC (Figure 3). This difference was statistically significant (t=-1.855; p=0.032). No significant differences in carcinoma incidence were observed between patients with benign FNA results and those who did not undergo FNA.

### Discussion

The observed incidence of 14.4% higlight a significant risk of thyroid carcinoma development in patients with MNG compared to the general population. This finding aligns with recent studies conducted in various Italian populations [14, 15], including those by Bove et al. (2023), Spaziani et al. (2023), and Chiefari et al. (2024) [3, 16, 6]. However, unlike these studies, which reported a significant prevalence in females, and the study by Apostolou et al. (2021) [4], which showed an increased incidence in males, our data revealed no notable sex-based differences in carcinoma distribution. This finding deviates from existing literature.

Although prevalence indices vary slightly, our findings regarding histotype distribution confirm, in agreement with numerous other studies [2-6, 15], that papillary thyroid carcinoma is the most prevalent subtype among patients with MNG, followed by follicular thyroid carcinoma.

It is noteworthy that Hurthle cell carcinoma, reported as such based on the 2018 histopathological classification, is now defined to as "oncocytic carcinoma" according to the 2022 WHO guidelines [18]. Given that half of the cases were papillary microcarcinomas, it is essential to emphasize their favorable prognosis despite their scientific interest. Although progression rates are below 15% over 10 years, they tend to increase with younger age at diagnosis [18, 19]. Older patients are ideal candidates for active surveillance with ultrasonographic monitoring, while younger patients may benefit more from surgery. However, most young patients would also qualify for active surveillance, as surgery may not be required during their lifetime [20, 21].

Regarding age as a risk factor for thyroid carcinoma in MNG patients, the literature reports conflicting data. Some studies found no significant relationship between age and malignancy [4, 22], whereas others, consistent with our findings, reported higher tumor prevalence in younger patients [23, 24]. Benign neoplasms, of which 22 cases were identified, require only conservative surgical management without the need for radioactive iodine therapy or ultrasonographic surveillance due to their low progression rates. Thyroid weight has been implicated as a potential risk factor for ITC [4, 22,

25,26,27]. Based on the existing literature [4, 22], clinical observations, and diagnostic pathways for malignancies in goitrous thyroids, we hypothesized that smaller thyroids with lower nodular density (cystic or spongiform appearance) are more prone to ITC, owing to diagnostic challenges with ultrasonography and FNA. This hypothesis was confirmed by our findings. Thyroid weight should therefore be considered a potential risk factor in the clinical management of MNG patients to ensure early detection of associated thyroid malignancies [28, 29].

The primary limitations of this study include the small sample size, the fact that the patients were recruited from a single center, and their representation of a genetically homogeneous population. While the latter reduces potential statistical errors related to genetic factors, it limits the generalizability of the findings.

The difficulty in collecting certain parameters due to incomplete data allowed for the evaluation of only a limited number of disease-related aspects, although these proved to be significant.

### Conclusion

The results of this study highlight a significant incidence of thyroid carcinoma in patients with multinodular goiter. The predominant histotype was papillary carcinoma, with no observed sex-based differences in incidence. The identified risk factors, such as age and thyroid weight, while potentially useful for stratifying risk in patients with multinodular goiter, are insufficient—due to study limitations and the significant variability among populations from different regions—to justify modifications to existing thyroid nodule screening criteria.

These results are an excellent starting point and instead underscore the need for multicenter studies aimed at developing specific monitoring protocols for this patient population. Such protocols could enable timely and targeted interventions, ultimately improving clinical outcomes and reducing morbidity associated with thyroid carcinoma.

## Bibliography

- 1. Pinchera A, Aghini-Lombardi F, Antonangeli L, Vitti P. Gozzo multinodulare. Epidemiologia e prevenzione [Multinodular goiter.
  - Epidemiology and prevention]. Ann Ital Chir. 1996 MayJun;67(3):317-25.
- 2. Campbell MJ, Seib CD, Candell L, Gosnell JE, Duh QY, Clark OH, Shen WT. The underestimated risk of cancer in patients with multinodular goiters after a benign fine needle aspiration. World J Surg. 2015 Mar;39(3):695-700.
- 3. Bove A, Manunzio R, Palone G, Di Renzo RM, Calabrese GV, Perpetuini D, Barone M, Chiarini S, Mucilli F. Incidence and Clinical Relevance of Incidental Papillary Carcinoma in Thyroidectomy for Multinodular Goiters. J Clin Med. 2023 Apr 7;12(8):2770.
- 4. Apostolou K, Zivaljevic V, Tausanovic K, Zoric G, Chelidonis G, Slijepcevic N, Jovanovic M, Paunovic I. Prevalence and risk factors for thyroid cancer in patients with multinodular goitre.

  BJS Open. 2021 Mar 5;5(2):zraa014.
- 5. Tartaglia N, Di Lascia A, Vovola F, Cianci P, Fersini A, Pacilli M, Pavone G, Ambrosi A. *Bilateral central neck dissection in the treatment of early unifocal papillary thyroid carcinomas with poor risk factors: A mono-institutional experience*. Ann Ital Chir. 2019 Dec 20;8. pii: S0003469X19031646. [Epub ahead of print]
- 6. Chiefari E, Innaro N, Gervasi R, Mirabelli M, Giuliano S, Donnici A, Obiso S, Brunetti FS, Foti DP, Brunetti A. Incidental thyroid carcinoma in an endemic goiter area in Italy: histopathological features and predictors of a common finding. Endocrine. 2024 May;84(2):589-597.
- 7. Kim K, Cho SW, Park YJ, Lee KE, Lee DW, Park SK. Association between Iodine Intake, Thyroid Function, and Papillary Thyroid Cancer: A Case-Control Study. Endocrinol Metab (Seoul). 2021 Aug;36(4):790-799.
- **8.** Zhao ZG, Guo XG, Ba CX, Wang W, Yang YY, Wang J, Cao HY. Overweight, obesity and thyroid cancer risk: a meta-analysis of cohort studies. J Int Med Res. 2012;40(6):2041-50.
- 9. Franchini F, Palatucci G, Colao A, Ungaro P, Macchia PE, Nettore IC. Obesity and Thyroid Cancer Risk: An Update. Int J Environ Res Public Health. 2022 Jan 20;19(3):1116.
- 10. Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM,

- Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133.
- Pacilli M, Tartaglia N, Gerundo A, Pavone G, Fersini A, Ambrosi A. Energy Based Vessel Sealing Devices in Thyroid Surgery: A Systematic Review to Clarify the Relationship with Recurrent Laryngeal Nerve Injuries. Medicina (Kaunas). 2020 Nov 27;56(12):651. doi: 10.3390/medicina56120651. PMID: 33260912; PMCID: PMC7760641.
- **12.** Al-Yaarubi S, Farhan H, Al-Futaisi A, Al-Qassabi S, Al-Rasadi K, AlRiyami S, Al-Zakwani I. Accuracy of ultrasound-guided fine-needle aspiration cytology for diagnosis of carcinoma in patients with multinodular goiter. Indian J Endocrinol Metab. 2011 Jul;15(Suppl 2):S132-5.
- 13. Nikiforov YE, Carty SE, Chiosea SI, Coyne C, Duvvuri U, Ferris RL, Gooding WE, LeBeau SO, Ohori NP, Seethala RR, Tublin ME, Yip L, Nikiforova MN. Impact of the Multi-Gene ThyroSeq NextGeneration Sequencing Assay on Cancer Diagnosis in Thyroid Nodules with Atypia of Undetermined Significance/Follicular Lesion of Undetermined Significance Cytology. Thyroid. 2015 Nov;25(11):1217-23.
- **14.** Cancer Genome Atlas Research Network. Integrated genomic characterization of papillary thyroid carcinoma. Cell. 2014 Oct 23;159(3):676-90.
- **15.** Costamagna D, Pagano L, Caputo M, Leutner M, Mercalli F, Alonzo A. Incidental cancer in patients surgically treated for benign thyroid disease. Our experience at a single institution. G Chir. 2013 JanFeb;34(1-2):21-6.
- **16.** Pezzolla A, Marzaioli R, Lattarulo S, Docimo G, Conzo G, Ciampolillo A, Barile G, Anelli FM, Madaro A. Incidental carcinoma of the thyroid. Int J Surg. 2014;12 Suppl 1:S98-102.
- 17. Spaziani E, Di Filippo AR, Di Cristofano C, Tamagnini GT, Spaziani M, Caruso G, Salina G, Valle G, Picchio M, De Cesare A. Incidental papillary thyroid microcarcinoma in consecutive patients undergoing thyroid surgery for benign disease. A single center experience. Ann Ital Chir. 2023;94:142-146.

- **18.** Baloch ZW, Asa SL, Barletta JA, Ghossein RA, Juhlin CC, Jung CK, LiVolsi VA, Papotti MG, Sobrinho-Simões M, Tallini G, Mete O. Overview of the 2022 WHO Classification of Thyroid Neoplasms. Endocr Pathol. 2022 Mar;33(1):27-63.
- 19. Pacilli M, Pavone G, Quazzico A, Fersini A, Ambrosi A, Tartaglia N. Ultrasound-guided approach to surgery for nodal recurrence following lateral neck dissection for differentiated thyroid carcinoma. A single institution experience. Front Surg. 2024 Jun 25;11:1403741. doi: 10.3389/fsurg.2024.1403741. PMID: 38983587; PMCID: PMC11231422.
- **20.** Nagaoka R, Ebina A, Toda K, Jikuzono T, Saitou M, Sen M, Kazusaka H, Matsui M, Yamada K, Mitani H, Sugitani I. Multifocality and Progression of Papillary Thyroid Microcarcinoma During Active Surveillance. World J Surg. 2021 Sep;45(9):2769-2776.
- 21. Miyauchi A, Kudo T, Ito Y, Oda H, Sasai H, Higashiyama T, Fukushima M, Masuoka H, Kihara M, Miya A. Estimation of the lifetime probability of disease progression of papillary microcarcinoma of the thyroid during active surveillance. Surgery.

  2018 Jan;163(1):48-52.
- 22. Sugitani I, Ito Y, Takeuchi D, Nakayama H, Masaki C, Shindo H, Teshima M, Horiguchi K, Yoshida Y, Kanai T, Hirokawa M, Hames KY, Tabei I, Miyauchi A. Indications and Strategy for Active Surveillance of Adult Low-Risk Papillary Thyroid Microcarcinoma: Consensus Statements from the Japan Association of Endocrine

  Surgery Task Force on Management for Papillary Thyroid Microcarcinoma. Thyroid. 2021 Feb;31(2):183-192.
- **23.** Ito Y, Miyauchi A. Active surveillance of low-risk papillary thyroid microcarcinomas. Gland Surg. 2020 Oct;9(5):1663-1673.
- 24. Pacilli M, Pavone G, Gerundo A, Fersini A, Ambrosi A, Tartaglia N. Clinical Usefulness of the Valsalva Manoeuvre to Improve Hemostasis during Thyroidectomy. J Clin Med. 2022 Sep 29;11(19):5791. doi: 10.3390/jcm11195791. PMID: 3623365
- **25.** Luo J, McManus C, Chen H, Sippel RS. Are there predictors of malignancy in patients with multinodular goiter? J Surg Res. 2012 May 15;174(2):207-10.
- **26.** Miccoli P, Minuto MN, Galleri D, D'Agostino J, Basolo F, Antonangeli L, Aghini-Lombardi F, Berti P. Incidental thyroid carcinoma in a large series of consecutive patients operated on for benign thyroid disease. ANZ J Surg. 2006 Mar;76(3):123-6.

- **27.** De Carlos J, Ernaga A, Irigaray A, Pineda JJ, Echegoyen A, Salvador P, Anda E. Incidentally discovered papillary thyroid microcarcinoma in patients undergoing thyroid surgery for benign disease. Endocrine. 2022 Aug;77(2):325-332.
- 28. Pacilli M, Tartaglia N, Pavone G, De Fazio M, Ambrosi A, Fersini A. Indocyanine green fluorescence angiography in parathyroidectomy for primary hyperparathyroidism. Ann Ital Chir. 2022;93:621-625. PMID: 36617270.
- 29. Erbil Y, Barbaros U, Salmaslioglu A, Mete O, Issever H, Ozarmagan S, Yilmazbayhan D, Tezelman S. Effect of thyroid gland volume in preoperative detection of suspected malignant thyroid nodules in a multinodular goiter. Arch Surg. 2008 Jun;143(6):558-63; discussion 563.